CLINICAL TRIAL: NCT06821672
Title: The Effect of Chronobiological Feeding Model on Sleep and Physiological Conditions of Neonates: A Randomized Controlled Study"
Brief Title: The Effect of Oral Feeding Model With a Chronobiological Approach in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, ebru temizsoy, PhD, RN, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/0161
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Preterm; Chronobiology; Human Milk/Breastfeeding; Bottle Feeding; Sleep Disorders, Circadian Rhythm
Keywords: preterm Human milk Circadian rhythm neonate, sleep, cry
MeSH Terms: conditions — Premature Birth; Bottle Feeding; Sleep Disorders, Circadian Rhythm; Crying

STUDY DESIGN:
Intervention Model Description: Randomized Controlled two groups (control group and study group)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No Intervention: Control Group Preterm infants in the NICU are fed with breast milk and bottles. Although the date is written on the expressed breast milk, it is usually not given after checking the time of day. The experiment is about labeling the breast milk according to the time of day before giving it to the babies. No extra intervention is made during feeding. The breast milk of the control group patients will be given without being matched according to the clinical routine practice. Demographic data, measurements of sleep characteristics (time and quality), and characteristics of physiological status will be recorded on the "Baby Monitoring Form" created by the researcher.
- Intervention Group (Experimental): Experimental: Chronobiological Approach Nutrition Model Preterm infants in NICU are fed with breast milk and bottle. Although the date is written on expressed breast milk, it is usually not given by checking its suitability for the time of day. The milk of the intervention group patients will be matched circadian and given to the babies. Intervention group's breast milk is labeling by time of day before the each feeding. In the intervention group, a label containing the time of expressed breastmilk will be affixed. Circadian matched milk will be provided at each feeding. intervention is;n the intervention group, a label containing the time of expressed breastmilk will be affixed. In the milk preparation room, breast milk will be stored in a separate refrigerator as 08:00-19:59 day milk and 20:00-07:59 night milk. Demographic data, measurements of sleep characteristics (duration and quality), and characteristics of physiological status will be recorded on the "Baby Monitoring Form"
  Interventions: Procedure: Chronobiological Group

INTERVENTIONS:
Procedure: Chronobiological Group — In the intervention group, a label containing the time of expressed breastmilk will be affixed. In the milk preparation room, breast milk will be stored in a separate refrigerator as 08:00-19:59 day milk and 20:00-07:59 night milk.
  Arms: Intervention Group

SUMMARY:
The ideal food for healthy term babies as well as preterm babies and sick term babies is breast milk. There are many studies showing that the composition of breast milk can vary from mother to mother, according to the baby's gestational age and gender. New studies on the content of breast milk suggest that breast milk is different during the day and at night, that micro and macronutrient content, hormones and some enzymes are secreted at different levels at different times of the day and that breast milk has a circadian rhythm.

This study was designed as a prospective, randomized, controlled study. The study will be conducted to evaluate the effect of the Chronobiological Approach Feeding Model application on the baby's sleep characteristics and physiological conditions in preterm babies hospitalized in the Neonatal Intensive Care Unit (NICU).

The simple randomization method will be used in the study and the babies will be divided into intervention (n=30) and control (n=30) groups. The study was conducted with 60 infants followed in the neonatal intensive care unit.

The milk of the intervention group patients will be given to the babies by matching them circadianly , while the milk of the control group patients will be given without matching according to clinical routine practice. Demographic data and sleep measurements (time and quality) of all infants will be recorded in the "Baby Monitoring Form" created by the researcher.

DETAILED DESCRIPTION:
Circadian fluctuations in breast milk content are very important in preterm infants fed with breast milk. The composition of breast milk changes throughout the day. There is no randomized controlled study in the literature suggesting that breast milk should be matched to the infant's circadian. This study aimed to evaluate the effect of the Chronobiological Nutrition Model application on the sleep characteristics and physiological conditions of preterm infants in the neonatal intensive care unit. It is aimed to increase the sleep duration and depth of infants, shorten the crying periods and increase the quality of nursing practices by circadian matching with breast milk in the feeding of preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants with family consent,
* 32 0/6 - 36 6/7 weeks of gestation,
* Exclusively breastfed,
* Infants who have switched to full oral feeding

Exclusion Criteria:

* Intravenous fluid therapy,
* Feeding intolerance
* Sepsis, Necrotizing enterocolitis, Major congenital anomaly,
* Mechanical ventilation support.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Sleep time | 24 hour
  Effect of Chronobiological Approach Feeding Model on infant sleep time during circadian matched breastfeeding sleep time in hours
Crying time | 24 hour
  Effect of Chronobiological Approach Feeding Model on infant crying duration measured during circadian matched breastfeeding crying duration in hours

SECONDARY OUTCOMES:
Discharge time | through study completion, an average of 30 days]
  The effect of Chronobiological Approach Nutrition Model application on infant's hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: ebru temizsoy, PhD, Principal Investigator — İstanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No